CLINICAL TRIAL: NCT05313061
Title: Effect of One-week Discontinuation of Methotrexate on Immunogenicity of COVID-19 Booster Vaccination in Patients With Rheumatoid Arthritis: A Randomized Pilot Study
Brief Title: MTX Hold During Covid-19 Booster
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2112-019-1279
Record Dates: First submitted 2021-12-28; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX continue (Active Comparator): Group will continue MTX after vaccination
  Interventions: Drug: MTX
- MTX 1 week hold (Experimental): Group will continue MTX for 1 week after vaccination
  Interventions: Drug: MTX

INTERVENTIONS:
Drug: MTX — MTX continuation

SUMMARY:
To investigate the effect of MTX discontinuation for 1 week on vaccination response to Covid-19 booster vaccination in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 19 years of age at time of consent
* Have a diagnosis of RA per ACR criteria
* Require methotrexate for RA treatment
* Subject to a Covid-19 booster vaccination
* Must understand and voluntarily sign an informed consent form including writing consent for data protection

Exclusion Criteria:

* Pregnant or lactating females
* Previous anaphylactic response to the vaccine components
* Any other rheumatic disease such as systemic lupus erythematosus, mixed connective tissue disease, dermatomyositis/polymyositis, and vasculitis except for secondary Sjogren's disease
* Any condition including laboratory abnormality which places the subject at unacceptable risk
* Subjects who decline to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Covid-19 antibody titer before and after Covid-19 vacciation | 2 weeks
  Titer and geometric mean titers (GMTs) of neurolizing antibody after vaccination

SECONDARY OUTCOMES:
T cell activation after vaccination | 2, 4, 16 weeks
  Percentage of activated T cells after vaccination
B cell activation after vaccination | 2, 4, 16 weeks
  Percentage of activated b cells after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JK, Lee YJ, Shin K, Ha YJ, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Impact of temporary methotrexate discontinuation for 2 weeks on immunogenicity of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2018 Jun;77(6):898-904. doi: 10.1136/annrheumdis-2018-213222. Epub 2018 Mar 23. PMID 29572291
- [Background] Park JK, Lee MA, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Effect of methotrexate discontinuation on efficacy of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2017 Sep;76(9):1559-1565. doi: 10.1136/annrheumdis-2017-211128. Epub 2017 May 3. PMID 28468794
- [Background] Curtis JR, Johnson SR, Anthony DD, Arasaratnam RJ, Baden LR, Bass AR, Calabrese C, Gravallese EM, Harpaz R, Kroger A, Sadun RE, Turner AS, Williams EA, Mikuls TR. American College of Rheumatology Guidance for COVID-19 Vaccination in Patients With Rheumatic and Musculoskeletal Diseases: Version 3. Arthritis Rheumatol. 2021 Oct;73(10):e60-e75. doi: 10.1002/art.41928. Epub 2021 Aug 4. PMID 34346564